CLINICAL TRIAL: NCT01855711
Title: A Four-week, Open, Multicenter Study to Assess the Safety and Efficacy of 1 mg Once Daily (QD) of GR68755 in Female Subjects With Severe Diarrhea-predominant Irritable Bowel Syndrome (IBS) Who Have Frequent Bowel Urgency
Brief Title: Safety and Efficacy Study of GR68755 (Alosetron Hydrochloride) to Treat Severe Diarrhea-Predominant Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S3B20032
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Irritable Colon
Keywords: Alosetron hydrochloride; Global Improvement Scale(GIS); Diarrhea-predominant IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alosetron; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GR68755 (Alosetron hydrochrolide) group (Experimental): GR68755 1 mg tablets QD in the morning every day for 28 days
  Interventions: Drug: GR68755 (Alosetron hydrochloride) 1 mg tablet

INTERVENTIONS:
Drug: GR68755 (Alosetron hydrochloride) 1 mg tablet — 1 tablet (1 mg) once a day

SUMMARY:
This study is an exploratory study aiming (i) to obtain clinical experience of GR68755 in Japanese subjects with severe d-IBS to explore the feasibility of the next phase study and (ii) to obtain reference data for endpoints and dosage and administration of a next phase study.

DETAILED DESCRIPTION:
The study objectives are to obtain the clinical experience of GR68755 1 mg QD in Japanese female subjects with severe d-IBS who have frequent bowel urgency and to obtain exploratory efficacy and safety data that can be used as reference for endpoints and dosage and administration of a next phase clinical study in Japan.

After giving a written informed consent, subjects will undergo essential observation and examinations during the screening phase and subjects who meet the eligibility criteria will enter into the treatment phase. When subjects enter into the treatment phase, the subjects will administer GR68755 1 mg tablets QD in the morning every day for 28 days from the next day of receiving the investigational products.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Disease to be treated: Has been diagnosed with severe d-IBS (at least 6 months of d-IBS symptoms as defined by the Rome II Criteria), and failed conventional IBS therapy.

   The following criteria (2. and 3.) will be confirmed at the end of screening phase (before assigning the investigational products) based on the record in the diary card.
2. Meets both (1) and (2) during the 1-week screening phase. (1)Has recorded symptom data on at least 6 days in the diary card during the screening phase. In case of patient whose screening phase is 5 days, has recorded symptom data on all days (5 days) in the diary card during the screening phase (2)An average stool consistency score recorded in the diary card during the screening phase is >=3.0.

Stool consistency score

1. = very hard
2. = hard
3. = formed
4. = loose
5. = watery 3.Meets both the following (1) and (2):

(1)Average "severity of abdominal pain or discomfort" score recorded in the diary card during the screening phase is >=1.0 (2)Has frequent "bowel urgency" (has urgency >= 50% of the days during the screening phase) Severity of pain or discomfort score

1. = mild
2. = moderate
3. = intense
4. = severe However, if the subject did not experience abdominal pain or discomfort, score zero (0).

4.Age: Is 20-64 years of age 5.Sex: Female 6.Type of subject: Outpatient 7.Is ambulatory (not depending on a wheelchair for mobility) 8.Is not pregnant, lactating, or intend to become pregnant during the study period.

Females of a non-child bearing potential are allowed to participate in this study if one of the following criteria are met:

-Sterilization (via hysterectomy or bilateral tubal ligation)

* Post-menopausal (is defined as one year without menses) Females of child-bearing potential may also be enrolled if they subject demonstrate a negative serum β-hCG test at the screening, and agree to practice contraception throughout the study. The following methods of contraception are acceptable.
* Oral birth control pills administered for at least one monthly cycle prior to the investigational product administration
* An IUD (intrauterine contraceptive device)
* Complete abstinence from intercourse for two weeks prior to the investigational product administration throughout the study period.

  9.Has normal results from the following tests and symptoms have remained stable, according to subject's age, within two years of the screening visit after IBS symptoms have developed.

<50 years of age: a sigmoidoscopy, a sigmoidoscopy plus barium enema, or a colonoscopy.

=>50 years of age: a sigmoidoscopy plus barium enema, or colonoscopy. If a subject has not performed a flexible sigmoidoscopy, flexible sigmoidoscopy plus barium enema, or colonoscopy after development of IBS and within 2 years of the screening visit, the appropriate procedure will be performed after being judged as eligible for this study during the procedure window. After completing the tests, at least three days interval should be provided before entering into the treatment phase. However, the maximum interval from the completion of the tests to the entry into the treatment phase is 7 days. If subject is not eligible based on the data recorded on the diary card until the day of above tests conducted, subject should withdraw the study prior to the tests.

10.Is able to give a written informed consent.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Does not have severe d-IBS
2. Has current evidence of or history of chronic or severe constipation, or a history of sequelae from constipation.
3. Is currently constipated or did report no stool for three or more consecutive days during the screening phase.
4. Has evidence of bloody diarrhea or abdominal pain with lower gastrointestinal hemorrhage.
5. Has current evidence of uncontrollable cardiovascular, renal, hepatic, pulmonary, endocrine, metabolic, hematologic, or digestive condition (excluding IBS).
6. Has evidence of biochemical or structural abnormality of the digestive tract.

   These conditions include the evidence or history of the following:
   * Ischemic colitis
   * Impaired intestinal circulation
   * gastrointestinal perforation
   * gastrointestinal obstruction and/or stricture
   * diverticulitis
   * Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
   * Microscopic colitis (lymphocytic colitis, collagenous colitis), or celiac sprue
   * Laxative abuse (in the clinical judgement of the investigator/subinvestigator) or melanosis coli.
   * Gastroparesis
   * GI malignancy
   * Carcinoid syndrome
   * Amyloidosis
   * Chronic pancreatitis
   * Abdominal adhesions
   * Toxic megacolon
   * Acute proctitis
   * Fecal impaction
   * Symptomatic cholelithiasis
7. Has performed gastrointestinal surgery (except six months post-surgery appendectomy, cholecystectomy, benign polypectomy, fundoplication (not have gas bloat), and hiatal hernia repair; three months post-surgery herniorrhaphy without bowel resection)
8. Has a history of thrombophlebitis or hypercoagulable state.
9. Has been diagnosed with a psychiatric disorder that required hospitalization and/or involved a suicide attempt (however, if a subject has a history of severe psychiatric disorder other than above within the past two years, the subject may enter into the study if the symptom is controlled with a stable dose of medicine for at least six months prior to the screening visit)
10. Has a history of alcohol and/or drug abuse within the past two years.
11. Exhibits evidence of hepatic dysfunction (AST [GOP] or ALT [GPT] values >2.5 times the upper limit of normal or alkaline phosphatase or serum bilirubin values >2.0 times the upper limit of normal)
12. Exhibits evidence of renal impairment (a serum creatinine value >2.0 mg/dl)
13. Exhibits an abnormal serum thyroid-stimulating hormone (TSH) (TSH value exceeds the limit of normal at the clinical laboratory).
14. Has current evidence of, or has been treated for a malignancy within the past five years (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected).
15. Has used GR68755 tablets or has been participated in other clinical study of 5HT3 antagonists in IBS patients within three years prior to the screening visit.
16. Has been enrolled in other clinical study within four months prior to the screening visit.
17. Has used any prohibited concomitant medicine within seven days prior to the screening visit. However loperamin hydrochloride and butylscopolamine bromide may be taken until 24 hours before starting the screening period.
18. Has used a permitted concomitant medication within 30 days prior to the screening visit and adjusted the dose.
19. Is hypersensitive to 5-HT3 antagonists.
20. Is pregnant or breastfeeding.
21. Is not eligible to participate this study in the opinion of the investigator/subinvestigator.

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2003-09-18 (Actual); Primary Completion 2005-05-10 (Actual); Study Completion 2005-05-10 (Actual)

PRIMARY OUTCOMES:
Global Improvement Scale(GIS) | four weeks
Satisfactory control of IBS related bowel urgency | four weeks

SECONDARY OUTCOMES:
Adequate relief of IBS pain and discomfort | four weeks
Days without abdominal pain and discomfort | four weeks
Severity score of abdominal pain and/or discomfort | four weeks
Intestine function(Number of bowel movement,Stool form,Feeling of incomplete evacuation,Abdominal bloating) | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline